CLINICAL TRIAL: NCT04756960
Title: Evaluation of the Absolute Bioavailability and Mass Balance of CHF6001 Following a Single Inhaled Dose Co-administered With an Intravenous Radiolabelled Microtracer Dose in Healthy Volunteers
Brief Title: Evaluation of the Absolute Bioavailability and Mass Balance of CHF6001 (Tanimilast) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLI-06001AA1-02; 2020-004201-31 (EudraCT Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Healthy subjects; Phase I; CHF6001; Tanimilast; Chiesi Farmaceutici S.p.A
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tanimilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHF6001 (Experimental): single dose of CHF6001 dry-powder inhaler (DPI) co-administered with an intravenous microdose of [14^C]-labelled CHF6001
  Interventions: Drug: CHF6001

INTERVENTIONS:
Drug: CHF6001 — 4 inhalations of CHF6001 800 µg/20 mg NEXThaler® dry-powder inhaler (DPI), (total dose of 3200µg) co-administered with an intravenous microdose (18.5µg (18.5 kBq)) of [14^C]-labelled CHF6001

SUMMARY:
The objective of the study is to evaluate the bioavailability of CHF6001 after inhaled administration, to characterize the mass balance and route of elimination of CHF6001 along with its relevant metabolites, in healthy male subjects.

DETAILED DESCRIPTION:
This clinical trial is a single centre Phase I study, with a single dose, non-randomized, open-label, uncontrolled design. A total of 8 healthy male subjects were included in the study.

The aim was to assess the absolute bioavailability, the mass balance, and routes of elimination of CHF6001 (Tanimilast) in healthy male subjects, using [14^C]-radiolabelled drug substance, administered as an intravenous (iv) infusion concomitantly with an inhaled (inh) non-radiolabelled dose of CHF6001.

Standard safety assessments were conducted during the study, including safety blood and urine laboratory tests, vital signs, physical examinations, ECGs, and assessment of any adverse events (AE). Blood, urine, and feces samples were collected for pharmacokinetic (PK) analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Able to understand the study procedures, the risks involved and ability to be trained to use correctly the inhalers and to generate sufficient Peak Inspiratory Flow (PIF), using the In-Check device and Placebo inhaler;
3. Male subjects aged 30 to 55 years inclusive;
4. Body mass index (BMI) within the range of 18 to 35 kg/m^2 inclusive;
5. Non- or ex-smoker who smoked < 5 pack years and who stopped smoking > 1 year prior to screening;
6. Good physical and mental status;
7. Vital signs at screening within limits;
8. 12-lead digitised Electrocardiogram (12-lead ECG) in triplicate considered as normal;
9. Lung function measurements within normal limits at screening;
10. Regular bowel movements at screening;
11. Males with non-pregnant Women of Childbearing Potential (WOCBP) partners: they and/or their partner of childbearing potential must be willing to use a highly effective birth control method in addition to the male condom from the signature of the informed consent and until 90 days after the follow-up visit. Males with pregnant WOCBP partner: they must be willing to use male contraception (condom) from the signature of the informed consent and until 90 days after the follow-up visit.

Exclusion Criteria:

1. Participation in another clinical trial with an investigational drug in the 3 months or 5 half-lives of that investigational drug (whichever is longer) preceding the administration of the study drug;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic (including Gilbert syndrome), gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorder;
3. Clinically relevant abnormal laboratory values;
4. Subjects with history of breathing problems;
5. Positive to Human Immunodeficiency Virus 1/Human Immunodeficiency Virus 2 (HIV1/HIV2) serology at screening;
6. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C at screening;
7. Blood donation or blood loss (equal or more than 450 mL) less than 2 months prior screening or prior to treatment;
8. Positive urine test for cotinine;
9. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test;
10. Documented history of drug abuse within 12 months prior to screening or a positive urine drug screen;
11. Intake of non-permitted concomitant medications in the predefined period;
12. Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or before treatment;
13. Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the trial;
14. Unsuitable veins for repeated venipuncture;
15. Heavy caffeine drinker;
16. Abnormal haemoglobin level at screening;
17. Subjects using e-cigarettes within 6 months prior to screening;
18. Subjects been involved in a study involving a 14^C-labeled drug within the 12 months prior to enrollment;
19. Subjects with exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to Day-1;
20. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 8 weeks or which has not resolved within 14 days prior to screening and before treatment.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance - Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CHF6001: Single dose of CHF6001 dry-powder inhaler (DPI) co-administered with an intravenous microdose of [14^C]-labelled CHF6001
  CHF6001: 4 inhalations of CHF6001 800µg/20mg NEXThaler® DPI (total dose of 3200µg) co-administered with an intravenous microdose (18.5µg (18.5kBq)) of [14^C]-labelled CHF6001
Period: Overall Study
Arm/Group | CHF6001
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Healthy male subjects.
Groups:
- CHF6001: Single dose of CHF6001 DPI co-administered with an intravenous microdose of [14^C]-labelled CHF6001
  CHF6001: 4 inhalations of CHF6001 800µg/20mg NEXThaler® DPI (total dose of 3200µg) co-administered with an intravenous microdose (18.5µg (18.5kBq)) of [14^C]-labelled CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.09 (4.73)

OUTCOME MEASURES:

1. Primary Outcome: PK Parameter -- AUC(0-t_iv) -- Plasma -- [14^C] Total
Description: AUC(0-t_iv) for [14^C] total in plasma.
  AUC(0-t_iv)=Area Under the curve, from 0 to the last quantifiable concentration, after intravenous (iv) infusion administration.
Time Frame: Pre-dose (within 60 min from inhaled dosing) and at the following timepoints relative to the start of the IV infusion: 5, 10, 15 [end of infusion], 20, 25, 30, 45, 60 min, 2, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours.
Population: Pharmacokinetic Population: all subjects from the safety population excluding subjects without any valid pharmacokinetic (PK) measurement or with major protocol deviations significantly affecting PK, for example: incorrect inhalation, change in subject condition (cold), failure in delivery of the device, use of non-permitted medications.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ngEq/mL
Groups:
- CHF6001: Single dose of CHF6001 DPI co-administered with an intravenous microdose of [14C]-labelled CHF6001
  CHF6001: 4 inhalations of CHF6001 800µg/20mg NEXThaler® DPI (total dose of 3200µg) co-administered with an intravenous microdose (18.5µg (18.5kBq)) of [14C]-labelled CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h*ngEq/mL | 5.4025 (16.7)

2. Primary Outcome: PK Parameter -- C(max_iv) -- Plasma -- [14^C] Total
Description: C(max_iv) for [14^C] total in plasma.
  C(max_iv)=Peak plasma concentration after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
ngEq/mL | 0.7072 (21.6)

3. Primary Outcome: PK Parameter -- t(max_iv) -- Plasma -- [14^C] Total
Description: t(max_iv) for [14^C] total.
  t(max_iv)=Time to reach the Cmax, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h | 0.217 [0.17 to 0.25]

4. Primary Outcome: PK Parameter -- AUC(0-∞_iv) -- Plasma -- [14^C] Total
Description: Area under curve extrapolated to infinity (AUC(0-∞_iv) for [14^C] total in plasma.
  AUC(0-∞_iv)=Area under curve extrapolated to infinity, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ngEq/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 6
h*ngEq/mL | 6.0825 (19.6)

5. Primary Outcome: PK Parameter -- t(1/2_iv) -- Plasma -- [14^C] Total
Description: Terminal half-life t(1/2_iv) for [14^C] total and CHF6001.
  t1/2_iv=Terminal half-life, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 6
h | 72.4057 [56.446 to 105.776]

6. Primary Outcome: PK Parameter -- (Blood to Plasma Ratio) -- Blood, Plasma -- [14^C] Total
Description: Blood to plasma ratio for [14^C] total.
Time Frame: Pre-dose (within 60 min from inhaled dosing) and at 20 min after the start of IV infusion.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | CHF6001
Number analyzed (Participants) | 6
Ratio | 0.6490 (23.9)

7. Primary Outcome: PK Parameter -- AUC(0-t_iv) -- Plasma -- [14^C] CHF6001
Description: AUC(0-t_iv) for [14^C] CHF6001 in plasma.
  AUC(0-t_iv)=Area Under the curve, from 0 to the last quantifiable concentration, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h*ng/mL | 0.7825 (18.2)

8. Primary Outcome: PK Parameter -- C(max_iv) -- Plasma -- [14^C] CHF6001
Description: C(max_iv) for [14^C] CHF6001 in plasma.
  C(max_iv)=Peak plasma concentration, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
ng/mL | 0.6312 (19.1)

9. Primary Outcome: PK Parameter -- t(max_iv) -- Plasma -- [14^C] CHF6001
Description: t(max_iv) for [14^C] CHF6001.
  t(max_iv)=Time to reach the Cmax, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h | 0.217 [0.17 to 0.25]

10. Primary Outcome: PK Parameter -- AUC(0-∞_iv) -- Plasma -- [14^C] CHF6001
Description: Area under curve extrapolated to infinity (AUC0-∞_iv) for [14^C] CHF6001 in plasma.
  AUC(0-∞_iv)=Area under curve extrapolated to infinity, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h*ng/mL | 0.8138 (18.6)

11. Primary Outcome: PK Parameter -- t(1/2_iv) -- Plasma -- [14^C] CHF6001
Description: Terminal half-life t(1/2_iv) for [14^C] CHF6001 in plasma.
  t(1/2_iv)=Terminal half-life, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h | 13.5816 [6.452 to 33.092]

12. Primary Outcome: PK Parameter -- Volume of Distribution During the Terminal Phase (Vz_iv) -- Plasma -- [14^C] CHF6001
Description: Volume of distribution during the terminal phase (Vz_iv) of [14^C] CHF6001 in plasma.
  Vz_iv=Volume of distribution during the terminal phase, after intravenous (iv) infusion administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Litres | 436.1078 (38.6)

13. Primary Outcome: PK Parameter -- Vdss_iv -- Plasma -- [14^C] CHF6001
Description: Vdss_iv=Volume of distribution is calculated at steady-state for [14^C] CHF6001 in plasma, after intravenous (iv) infusion administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Litres | 201.2514 (36.2)

14. Primary Outcome: PK Parameter -- Clearance (CL_iv) -- Plasma -- [14^C] CHF6001
Description: Systemic plasma clearance for [14^C] CHF6001.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres/h
Groups:
- CHF6001: Single dose of CHF6001 DPI co-administered with an intravenous microdose of [14C]-labelled CHF6001.
  CHF6001: 4 inhalations of CHF6001 800µg/20mg NEXThaler® DPI (total dose of 3200µg) co-administered with an intravenous microdose (18.5µg (18.5kBq)) of [14C]-labelled CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Litres/h | 21.9951 (18.6)

15. Primary Outcome: PK Parameter -- Blood to Plasma Ratio -- Blood, Plasma -- [14^C] CHF6001
Description: Blood to plasma ratio for [14^C] CHF6001.
Time Frame: Pre-dose (within 60 min from inhaled dosing) and at 20 min after the start of IV infusion.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | CHF6001
Number analyzed (Participants) | 6
Ratio | 0.5166 (54.9)

16. Primary Outcome: PK Parameter -- AUC(0-t)_inh -- Plasma -- CHF6001
Description: AUC(0-t)_inh for CHF6001 in plasma.
  AUC(0-t)_inh=Area Under the curve, from 0 to the last quantifiable concentration after inhalation of CHF6001
Time Frame: At baseline (pre-dose) (within 60 min from inhaled dosing) and at the following timepoints post inhaled dose: 15, 30, 60, 90 min, 2, 3.75, 5.75, 7.75, 9.75, 11.75, 13.75, 25.75, 49.75, 73.75, 97.75, 121.75, 145.75, 169.75, 193.75, 217.75, and 241.75 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h*pg/mL | 71088 (28.2)

17. Primary Outcome: PK Parameter -- C(max_inh) -- Plasma -- CHF6001
Description: C(max_inh) for CHF6001 in plasma.
  C(max_inh)=Peak plasma concentration after inhalation of CHF6001
Time Frame: Pre-dose (within 60 min from inhaled dosing) and at the following timepoints post inhaled dose: 15, 30, 60, 90 min, 2, 3.75, 5.75, 7.75, 9.75, 11.75, 13.75, 25.75, 49.75, 73.75, 97.75, 121.75, 145.75, 169.75, 193.75, 217.75, and 241.75 hours.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
pg/mL | 1979 (22.5)

18. Primary Outcome: PK Parameter -- t(max_inh) -- Plasma -- CHF6001
Description: t(max_inh) for CHF6001 in plasma.
  t(max_inh)=Time to reach the Cmax after inhalation of CHF6001
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h | 2.008 [2.00 to 3.75]

19. Primary Outcome: PK Parameter -- AUC(0-∞_inh) -- Plasma -- CHF6001
Description: AUC(0-∞_inh) for CHF6001 in plasma.
  AUC(0-∞_inh)=Area under curve extrapolated to infinity after inhalation of CHF6001
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h*pg/mL | 72403 (28.4)

20. Primary Outcome: PK Parameter -- t(1/2_inh) -- Plasma -- CHF6001
Description: t(1/2_inh) for CHF6001 in plasma.
  t(1/2_inh)=Terminal half-life, after inhalation of CHF6001
Time Frame: as for outcome 17
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | CHF6001
Number analyzed (Participants) | 8
h | 41.5691 [25.930 to 45.159]

21. Primary Outcome: PK Parameter -- Absolute Inhaled Bioavailability (F_inh) -- Plasma -- CHF6001
Description: Absolute inhaled bioavailability for CHF6001.
  F_inh=Inhaled absolute bioavailability based on AUC(0-∞) after inhalation of CHF6001 F_inh=(AUC(0-∞)_inh x Dose_iv)/ (AUC(0-∞)_iv x Dose_inh).
Time Frame: as for outcome 16
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Ratio | 0.4977 (26.8)

22. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Urine -- [14^C] Total
Description: Urine excreted fraction for cumulative [14^C] total.
Time Frame: Baseline (pre dose, -12-0h) and relative to the start of the IV infusion at: 0-4h, 4-8h, 8-12h, 12-24h, 24-48h, 48-72h, 72-96h, 96-120h, 120-144h, 144-168h, 168-192h, 192-216h, and 216-240h.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cumulative % of dose excreted in urine
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Cumulative % of dose excreted in urine
  0-4 h | 1.99 (0.523)
  4-8 h | 3.26 (0.552)
  8-12 h | 3.93 (0.549)
  12-24 h | 5.24 (0.554)
  24-48 h | 6.77 (0.519)
  48-72 h | 7.35 (0.553)
  72-96 h | 7.64 (0.622)
  96-120 h | 7.80 (0.673)
  120-144 h | 7.89 (0.703)
  144-168 h | 7.96 (0.720)
  168-192 h | 8.01 (0.729)
  192-216 h | 8.06 (0.763)
  216-240 h | 8.10 (0.771)

23. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Urine -- [14^C]-CHF6001
Description: Urine excreted fraction for cumulative [14^C]-CHF6001.
  Measurements in urine were performed. All measured values were below the limit of quantification of the bioanalytical method.
Time Frame: as for outcome 22
Population: Pharmacokinetic Population: all subjects from the safety population excluding subjects without any valid pharmacokinetic (PK) measurement or with major protocol deviations significantly affecting PK, for example: incorrect inhalation, change in subject condition (cold), failure in delivery of the device, use of non-permitted medications.
  Measurements in urine were performed and no substance was detected.
Measure: Mean (Standard Deviation); unit: (%) percent of injected [14C]-CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
(%) percent of injected [14C]-CHF6001
  0-4 h | 0.00 (0.00)
  0-8 h | 0.00 (0.00)
  0-12 h | 0.00 (0.00)
  0-24 h | 0.00 (0.00)
  0-48 h | 0.00 (0.00)
  0-72 h | 0.00 (0.00)
  0-96 h | 0.00 (0.00)
  0-120 h | 0.00 (0.00)
  0-144 h | 0.00 (0.00)
  0-168 h | 0.00 (0.00)
  0-192 h | 0.00 (0.00)
  0-216 h | 0.00 (0.00)
  0-240 h | 0.00 (0.00)

24. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Fecal -- [14^C] Total
Description: Fecal excreted fraction for cumulative [14^C] total.
Time Frame: Baseline (pre dose, Day -1) and relative to the start of the IV infusion at: 0-24h, 24-48h, 48-72h, 72-96h, 96-120h, 120-144h, 144-168h, 168-192h, 192-216h, and 216 -240h.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cumulative % of dose excreted in feces
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Cumulative % of dose excreted in feces
  0-24 h | 7.64 (12.0)
  24-48 h: number analyzed (Participants) | 7
  24-48 h | 38.9 (20.6)
  48-72 h: number analyzed (Participants) | 7
  48-72 h | 57.7 (8.53)
  72-96 h: number analyzed (Participants) | 7
  72-96 h | 64.9 (4.26)
  96-120 h | 68.6 (2.35)
  120-144 h | 69.6 (2.08)
  144-168 h: number analyzed (Participants) | 6
  144-168 h | 70.0 (2.09)
  168-192 h | 70.5 (2.19)
  192-216 h | 70.7 (2.22)
  216-240 h: number analyzed (Participants) | 7
  216-240 h | 70.8 (2.26)

25. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Fecal -- [14^C]-CHF6001
Description: Fecal excreted fraction for cumulative [14^C]-CHF6001.
Time Frame: as for outcome 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (%) percent of injected [14C]-CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
(%) percent of injected [14C]-CHF6001
  0-24 h | 0.0435 (0.0676)
  0-48 h | 0.1748 (0.0895)
  0-72 h | 0.2507 (0.0855)
  0-96 h | 0.2816 (0.0685)
  0-120 h | 0.3048 (0.0660)
  0-144 h | 0.3060 (0.0642)
  0-168 h | 0.3060 (0.0642)
  0-192 h | 0.3060 (0.0642)
  0-216 h | 0.3060 (0.0642)
  0-240 h | 0.3060 (0.0642)

26. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Urine and Fecal -- [14^C] Total
Description: Urine and fecal excreted fraction for cumulative [14^C] total.
Time Frame: Over 240 h after administration; please see timepoints for outcome #22 (urine) and #24 (fecal).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cumulative % of dose excreted
Arm/Group | CHF6001
Number analyzed (Participants) | 8
Cumulative % of dose excreted
  0-4 h | 1.99 (0.523)
  4-8 h | 3.26 (0.552)
  8-12 h | 3.93 (0.549)
  12-24 h | 12.9 (12.3)
  24-48 h | 45.6 (20.8)
  48-72 h | 65.1 (8.67)
  72-96 h | 72.5 (4.12)
  96-120 h | 76.4 (2.46)
  120-144 h | 77.5 (2.23)
  144-168 h | 77.9 (2.32)
  168-192 h | 78.5 (2.46)
  192-216 h | 78.7 (2.51)
  216-240 h | 78.9 (2.58)

27. Primary Outcome: PK Parameter -- Cumulative Excreted Fraction (in %) -- Urine and Fecal -- [14^C]-CHF6001
Description: Urine and Fecal excreted fraction for cumulative [14^C]-CHF6001.
Time Frame: Over 240 h after administration; please see timepoints for outcome #22 (urine) and #24 (fecal).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (%) percent of injected [14C]-CHF6001
Arm/Group | CHF6001
Number analyzed (Participants) | 8
(%) percent of injected [14C]-CHF6001
  0-24 h | 0.0435 (0.0676)
  0-48 h | 0.1748 (0.0895)
  0-72 h | 0.2507 (0.0855)
  0-96 h | 0.2816 (0.0685)
  0-120 h | 0.3048 (0.0660)
  0-144 h | 0.3060 (0.0642)
  0-168 h | 0.3060 (0.0642)
  0-192 h | 0.3060 (0.0642)
  0-216 h | 0.3060 (0.0642)
  0-240 h | 0.3060 (0.0642)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of the Informed Consent signature (screening visit at 31 to 3 days before the study treatment administration) until the subject's study participation ended (follow-up phone call or visit at 7 to 10 days after discharge or premature discontinuation).
Arm/Group | CHF6001
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF6001 (N=8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator should inform Chiesi Farmaceutici S.p.A. before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation.

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT04756960/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04756960/SAP_001.pdf